CLINICAL TRIAL: NCT05816135
Title: Investigation of Environmental Parameters in Operating Rooms and Their Association With Surgical Site Infections During Orthopedic Implant Related Surgeries.
Brief Title: Investigation of Environmental Parameters in Operating Rooms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Getinge Group (Other)
Responsible Party: Principal Investigator, Maziar Mohaddes Ardebili, Professor, Sahlgrenska University Hospital
Other Study IDs: Getinge study
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Surgical Site Infection
Keywords: Colony forming units; Particles; Environmental parameters; Operating room; Surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative surgical site infection (SSI) is a serious and complicated healthcare-associated infection (HAI) affecting about 2% of patients undergoing orthopedic surgery. Exogenous infections, could occur from insufficient air quality in operating rooms as shown in previous studies. However, from our knowledge, no study have collect environmental parameters and cross referenced the data with recorded patient registries to see if insufficient air quality is associated with higher risk of exogenous SSI. Temperature, humidity and the difference in air pressure in relation to the operating room and the adjacent corridors are examples of environmental parameters that could affect the air quality in operating rooms. Number of persons during an operation and particle counts could also give an indication of insufficient air quality.

DETAILED DESCRIPTION:
Postoperative surgical site infection (SSI) is a serious and complicated healthcare-associated infection (HAI) affecting about 2% of patients undergoing orthopedic surgery. The source of the SSI can be the patient's own bacteria, which have entered the wound e.g. via the bloodstream or the skin, giving rise to so called endogenous infection. Exogenous infection is instead when the wound is contaminated from an external source, e.g. from skin particles shredded from the operating personnel or from other airborne bacterial- containing particles that end up directly in the wound of the patient. The particles can also fall on surfaces causing indirect wound contamination via surgical instruments or via the surgeon's hands. The consequences of SSI are usually greatest when a foreign body, such as an implant, has been placed into the patient's body. The foreign material gives the bacteria a surface to attach to and to form biofilm on, which protects the bacteria against both the body's immune system and antibiotic treatment.

In 2019, approximately 19,000 hip prostheses and 15,000 knee prostheses surgeries were performed in Sweden. The consequences of a prosthetic infection for the patient include longer care and rehabilitation time, long-term pain, risk of reoperation, and increased mortality. An especially vulnerable group is the elderly, fragile patients, who are more susceptible to getting an infection and are most likely to have a mortal outcome.

SSI after orthopedic implant-related surgery also has economic consequences for the healthcare, with an extra cost of 0.5-1 MSEK/deep infection. Based on these socio-economic and humane reasons, there is a great need to prevent SSI. Another reason is the increasing development of antibiotic resistance, which threatens the possibilities of effectively preventing and treating SSI.

Airborne contamination is considered a very important exogenous source of infection. In a land-mark study from 1982 it was showed that ultraclean air in operating rooms (< 10 bacteria-carrying particles (CFU)/m3) reduced the incidence of deep sepsis by 1/3 after total joint-replacement operations compared with control- operating rooms. In addition, there was a substantial reduction in the mean numbers of bacteria isolated from wounds during operations performed under ultraclean-air conditions compared with those isolated from wounds during operations in the control rooms.

In a previous study, we are addressing the issue of possible relationship between air contamination - measured as colony forming units (CFU)/m3, bacteria present in the wound, and the occurrence of SSI. In the study, the bacteriological findings and the incidence of SSI are evaluated in relation to conventional ventilated operating rooms and conventional ventilated operating rooms with the addition of local clean airflow over the surgical instruments. Because particles in the air act as means of transportation for bacteria, there is a consensus that the risk of bacterial airborne infection can be prevented by keeping particle levels as low as possible in the operating room. The most obvious way of controlling the number of particles in the air is via ventilation. The most common types of ventilation in an operating room today is mixed ventilation (also called displaced or conventional ventilation) or vertical laminar airflow (LAF). However, both these systems are very sensitive to disturbances of the airflow caused by e.g. door openings, the number of staff working inside the room and their movements and obstructive objects, as shown in previous studies.

The golden standard of microbial surveillance today is via measuring CFU during on going surgery. This gives a good estimation of bacteria in the operating room. However, the method is time and resource consuming, and requires handling of microbial sampling and incubation. As incubation takes approximately 2 days, the results are delivered to late before any intervention could be made. Particle counting could be used as a proxy-unit instead of CFU to give an indication of microbial presence in real-time. However, the association between CFU and particles must be investigated further for such an assumption to be made.

Environmental factors such as temperature, humidity and the difference in air pressure in relation to the operating room and the adjacent corridors also affect the air quality in operating rooms. The significance of these factors for bacterial airborne infection is, so far, relatively unknown and unexplored field of research and therefore of interest to investigate further.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic implant related surgery
* Surgery in operating rooms with installed equipment

Exclusion Criteria:

* Non-implant related surgery
* No Swedish citizen (no personal-id number)
* Revision surgery due to infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects included in the study are patients who are getting either arthroplasty surgery or fixation with nails and/or plates due to fracture or arthritis. Patients who are going through a revision surgery are also included, with the exception of revision due to infection.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of bacteria (CFU) and particles | 02/28/2022 - 06/31/2023
  By measuring particles and CFU in proximity of each other, an association between the two units can be used to predict the CFU, based on the particle count.
Environmental parameters association with surgical site infections | 01/01/2021 - 12/31/2023
  Environmental parameters (temperature, humidity, air pressure, door openings, persons present, particles) are being recorded into a database and cross referenced with patient registries to investigate the association with surgical site infections

CONTACTS AND LOCATIONS:
Overall Officials: Maziar Mohaddes, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden